CLINICAL TRIAL: NCT06204406
Title: A Multicenter, Prospective, Observational Clinical Study to Evaluate the Prognosis of Patients With Upper Tract Urothelial Carcinoma Receiving Kidney-sparing Therapy
Brief Title: Prognosis of Patients With Upper Tract Urothelial Carcinoma Receiving Kidney-sparing Therapy
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Tianjin Medical University Second Hospital (Other); Xiangya Hospital of Central South University (Other); West China Hospital (Other); Ruijin Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); The Second Hospital of Anhui Medical University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-081-B
Record Dates: First submitted 2023-11-26; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Upper Tract Urothelial Carcinoma Receiving Kidney-sparing Therapy
Keywords: kidney-sparing therapy; upper tract urothelial carcinoma
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with non-metastatic upper tract urothelial carcinoma receiving kidney-sparing therapy: The enrolled patients were patients with limited-stage or locally advanced UTUC, who were classified into the following four categories according to the 2022 EAU guidelines as low-risk and high-risk: 1) low-risk patients who were willing to undergo kidney-sparing surgery directly; 2) High-risk patients, with solitary kidney, functional single kidney, bilateral tumors, and absolute kidney-sparing indications; 3) High-risk patients with renal insufficiency, or diseases that lead to renal insufficiency, have relative indications for kidney protection; 4) High-risk patients with good renal function, but a particularly strong willingness to preserve the kidney, willing to accept clinical studies and participate in kidney preservation.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is a prospective observational study with observation only and no intervention

SUMMARY:
Upper tract urothelial carcinoma (UTUC) is a rare malignant disease which accounts for 5-10% of urothelial carcinoma in the western world and 9%-30% in China. About two thirds of patients have muscle invasive disease at diagnosis. Those patients usually have poor prognosis. The 5 year cancer specific survival is <50% for pT2/T3 and <10% for pT4. Radical nephroureterectomy is the standardized treatment for non-metastatic high risk UTUC. However, about half patients may suffer from impaired renal function after nephroureterectomy. On the other hand, kidney sparing surgery can avoid renal function impairment, but the therapy is only recommended for few patients with low-risk disease. The treatment for urothelial carcinoma has changed rapidly in the past few years. Immune checkpoint inhibitors and novel agents such as ADCs have shown promising therapeutic effect and were approved for patients with metastatic UTUC. Meanwhile, a recent study shows that patients with high-risk disease can also receive kidney sparing surgery without compromising cancer specific survival and overall survival. This prospective, observational study aims to evaluate the prognosis of contemporary kidney sparing surgery in patients with UTUC with or without perioperative therapy in the real world.

DETAILED DESCRIPTION:
The patients that meet the Inclusion and Exclusion Criteria will enroll into this observational trial. The therapeutic schedule is purposed to spare the kidney of non-metastatic primary UTUC patients.

ELIGIBILITY:
Minimum Age: 18 Years Maximum Age: 90 Years Sex: All Gender Based: No Accepts Healthy Volunteers: No

Criteria:

Inclusion Criteria:

1. Histopathological confirmed upper tract urothelial carcinoma;
2. Refused radical nephroureterectomy, or eligible for the indications of kidney-sparing surgery;
3. Participants must be willing to attend the follow-up visits;
4. Sign informed consent.

Exclusion Criteria:

1. Unable to undergo kidney-sparing surgery;
2. Life expectancy < 6 months;
3. Previous anti-tumor therapy against UTUC, including systemic chemotherapy, surgery, radiotherapy, or immunotherapy identifying by investigators.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with non-metastatic upper tract urothelial carcinoma receiving kidney-sparing therapy
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Two-year events-free survival rate | Up to 2 years
  events-free survival defined as time from initiation of first protocol therapy until the first time to develop any local recurrence (local/bladder), distant metastases or any cause-related death.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  defined as time from initiation for protocol therapy to death.
Metastasis free surviva | Up to 2 years
  metastasis free survival defined as time from initiation of protocol therapy until the development of distal metastasis or death

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  The adverse events are evaluated per Common Terminology Criteria for Adverse Events (CTCAE) 5.0..

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No